CLINICAL TRIAL: NCT00354094
Title: A Phase 2B Long-Term, Randomized, Open-Label, Safety And Tolerability Trial Comparing [S,S]-Reboxetine (PNU-165442g) With Routine Care In Patients With Postherpetic Neuralgia (PHN).
Brief Title: [S,S]-Reboxetine Long Term Safety Study In Post-Shingles Pain.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to business/operational issues.
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6061030
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2007-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — O-methyl reboxetine

INTERVENTIONS:
Drug: [S,S]-Reboxetine

SUMMARY:
The purpose of this study is to assess the long term (up to 2 years) safety and tolerability of [S,S]-Reboxetine in patients with pain after shingles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pain present for more than 3 months after healing of the shingles skin rash.
* Patients at screening must have a score of >/=40mm on the pain visual analogue scale.

Exclusion Criteria:

* Patients with significant hepatic impairment.
* Patients with other severe pain, that may impair the self-assessment of pain due to postherpetic neuralgia (pain after shingles).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2006-11; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Vital signs
Physical examination
12-lead ECG
Hematology/Biochemistry
Adverse events

SECONDARY OUTCOMES:
Pain Visual Analogue Scale
Patient Global Impression of Change
Neuropathic Pain Symptom Inventory
Modified Brief Pain Inventory - Short Form
SF-12 Health Survey
EQ-5D
Analgesic Treatment Satisfaction Scale
Pain-related Medication Utilization

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (6):
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, San Antonio, Texas
- Argentina (2):
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
- Canada (3):
  - Pfizer Investigational Site, Greater Sudbury, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Chile (2):
  - Pfizer Investigational Site, Viña del Mar, Región de Valparaíso
  - Pfizer Investigational Site, Santiago, RM
- Pfizer Investigational Site, Split, Croatia
- India (6):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradhesh
  - Pfizer Investigational Site, Chandigarh, Punjab
  - Pfizer Investigational Site, Bangalore
  - Pfizer Investigational Site, Chennai
  - Pfizer Investigational Site, Hyderabad
  - Pfizer Investigational Site, New Delhi
- Lithuania (4):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Klaipėda
  - Pfizer Investigational Site, Panevezys
  - Pfizer Investigational Site, Šiauliai
- Pfizer Investigational Site, Mérida, Yucatán, Mexico
- Pfizer Investigational Site, Sopot, Poland
- Pfizer Investigational Site, Ourense, OURENSE, Spain
- Pfizer Investigational Site, Stockholm, Sweden
- United Kingdom (5):
  - Pfizer Investigational Site, Bexhill-on-Sea, East Sussex
  - Pfizer Investigational Site, Addlestone, SURREY
  - Pfizer Investigational Site, Alcester
  - Pfizer Investigational Site, East Sussex
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061030&StudyName=%5BS%2CS%5D-Reboxetine%20Long%20Term%20Safety%20Study%20In%20Post-Shingles%20Pain.